CLINICAL TRIAL: NCT01530594
Title: Lenalidomide and Low Dose Dexamethasone Versus Bortezomib, Lenalidomide and Low Dose Dexamethasone for Induction, in Patients With Previously Untreated Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2081-113
Record Dates: First submitted 2012-01-23; First posted 2012-02-10 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2012-02

CONDITIONS: Multiple Myeloma
Keywords: Untreated; Without intent for immediate autologous stem cell transplant
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Lenalidomide

ARMS (2):
- Lenalidomide (Active Comparator): Lenalidomide/Low dose Dex (LLD)
  Interventions: Drug: Lenalidomide/Low dose Dex; Drug: Lenalidomide
- Bortezomib/Lenalidomide (Experimental): Bortezomib/Lenalidomide/ Low dose Dex (BLLD)
  Interventions: Drug: Bortezomib/Lenalidomide/ Low dose Dex

INTERVENTIONS:
Drug: Lenalidomide/Low dose Dex — Lenalidomide/Low dose Dex (LLD)
  Arms: Lenalidomide
Drug: Bortezomib/Lenalidomide/ Low dose Dex — Bortezomib/Lenalidomide/ Low dose Dex (BLLD)
  Arms: Bortezomib/Lenalidomide
Drug: Lenalidomide — Lenalidomide/Low dose Dex (LLD
  Arms: Lenalidomide

SUMMARY:
This is a randomized phase III trial of CC-5013 (lenalidomide, NSC-703813) and low dose dexamethasone (LLD) versus bortezomib (PS-341, NSC-681239), lenalidomide and low dose dexamethasone (BLLD) for induction, in patients with previously untreated multiple myeloma without an intent for immediate autologous stem cell transplant.

ELIGIBILITY:
1. Patients must have newly diagnosed multiple myeloma
2. Patients must have received no prior chemotherapy for this disease. Patients must have received no prior radiotherapy to a large area of the pelvis (more than half of the pelvis). Prior steroid treatment is allowed provided treatment was not more than 2 weeks in duration. Patients must not have received any prior treatment with bortezomib or lenalidomide.
3. Patients must be ≥ 18 years of age at the time of registration.
4. Patients must have a Zubrod Performance Status (PS) of 0 - 3
5. Patients must have adequate marrow function as defined herein:
6. Platelet count ≥ 80 x 103/mcL,
7. ANC ≥ 1 x 103/mcL, and Hemoglobin (including patients who have been either transfused or treated with EPO) ≥ 9 g/dL.
8. Institutions must submit a local cytogenetics report and FISH analysis report
9. Patients with pathologic fractures, pneumonia at diagnosis or symptomatic hyperviscosity.
10. Patients must have a calculated or measured creatinine clearance > 30 cc/min.
11. Patients must not have uncontrolled, active infection requiring intravenous antibiotics
12. Patients must not have any psychiatric illness
13. Patients must not be Hepatitis B, Hepatitis C or HIV positive
14. Patients must not have a history of cerebral vascular accident with persistent neurologic deficits.
15. Patients must be able to take aspirin 325 mg daily
16. Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test
17. No prior malignancy is allowed except for adequately treated basal cell (or squamous cell) skin cancer, in situ cervical cancer or other cancer for which the patient has been disease-free for five years.
18. Patients must be offered participation in GEP molecular studies for the evaluation of genetic polymorphisms.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2009-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
comparison progression-free survival (PFS) in patients with newly diagnosed myeloma treated with lenalidomide plus low dose dexamethasone versus bortezomib plus lenalidomide and low dose dexamethasone | Four years

CONTACTS AND LOCATIONS:
Locations (1):
- King Faisal Specialist Hospital &Reseach Center, Riyadh, Saudi Arabia